CLINICAL TRIAL: NCT05281718
Title: An in Vitro Pilot Study of the Role of Factor IX as an Alternative to Bypassing Agents in the Treatment of Breakthrough Bleeds in Patients With Hemophilia A and Inhibitors Treated With Emicizumab.
Brief Title: Factor IX as Adjunctive Therapy to Emicizumab (EMIX)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-200
Record Dates: First submitted 2022-02-11; First posted 2022-03-16 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia A
Keywords: Hemophilia A with inhibitors; In vitro; Emicizumab
MeSH Terms: conditions — Hemophilia A | interventions — Factor IX

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient Group (Experimental): In vitro spiking experiments will be realized in plasmas from patients with severe haemophilia A on emicizumab using increasing concentrations of factor IX (rFIX), Activated prothrombin complex (aPCC) and recombinant VIIa (rFVIIa).
  Interventions: Drug: Factor IX

INTERVENTIONS:
Drug: Factor IX — Factor IX is on of the substrates of emicizumab.

SUMMARY:
This trial will enroll patients with severe hemophilia A. Experiments will be run in vitro by spiking patients' blood with different molecules (currently used and theoretically proposed as adjunctive therapy to emicizumab), therefore no more than minimal direct risk to patients is expected. This is a pilot preclinical study.

DETAILED DESCRIPTION:
The study aims to determine the hemostatic effect of different Factor IX (FIX) concentrates when added to the plasma of patients on emicizumab prophylaxis and compare it to the hemostatic effect obtained with the addition of bypassing agents (activated prothrombin complex aPCC, and recombinant VIIa rVIIA, recombinant porcine FVIII).

The investigators will study the hemostatic effect using Thrombin Generation assay (CAT) in the presence of different concentrations of FIX concentrates. The investigators will compare the hemostatic effect of added FIX to the effect of added bypassing agents (activated prothrombin complex aPCC, and recombinant VIIa rVIIA, recombinant porcine FVIII)

Plasma will be collected from patients with hemophilia A and inhibitors treated with Emicizumab, a group of plasma samples will be spiked with different concentrations of Factor IX. Thrombin generation profiles will be obtained using CAT.

Another group of plasma samples will be spiked with different concentrations of by passing agents (activated prothrombin complex aPCC, and recombinant VIIa rVIIA, recombinant porcine FVIII). Thrombin generation profiles will be obtained using CAT.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent/Assent Form
* Male patients, Age 12 years and older at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Diagnosis of severe hemophilia A and are receiving emicizumab prophylaxis, on a weekly maintenance regimen

Exclusion Criteria:

* Not able to sign consent
* Not willing to provide extra blood for the experiments.
* Patients carrying the diagnoses of other coagulopathies in addition to hemophilia A
* Patients that have received any hemostatic agent within 5 half-lives of the blood draw. This applies to any agent that might have been used for any reason prior to the blood draw and might affect the global hemostasis.

Ages: 12 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Determine the homeostatic effect of adding Factor IX concentrate to the plasma of patients with Hemophilia A with inhibitors on emicizumab using peak thrombin | 1 Year
  Peak thrombin is a thrombin generation profile. The investigators will compare the peak thrombin obtained when spiking patient's plasma with Factor IX concentrates to that obtained when spiking patient's plasma with aPCC and rFVIIa on emicizumab prophylaxis.
Determine the hemostatic effect of Factor IX concentrates and recombinant porcine FVIII when added to the plasma of patients with Hemophilia A with inhibitors on emicizumab using peak thrombin | 1 Year
  The investigators will compare the peak thrombin obtained when spiking patient's plasma with Factor IX concentrates to that obtained when spiking patient's plasma with recombinant porcine FVIII on emicizumab prophylaxis.
Determine the homeostatic effect of adding Factor IX concentrate to the plasma of patients with Hemophilia A with inhibitors on emicizumab using Endogenous Thrombin Potential (ETP) | 1 Year
  Endogenous Thrombin Potential is a thrombin generation profile. The investigators will compare the Endogenous Thrombin Potential obtained when spiking patient's plasma with Factor IX concentrates to that obtained when spiking patient's plasma with aPCC and rFVIIa on emicizumab prophylaxis.
Determine the hemostatic effect of Factor IX concentrates and recombinant porcine FVIII when added to the plasma of patients with Hemophilia A with inhibitors on emicizumab using Endogenous Thrombin Potential (ETP) | 1 Year
  The investigators will compare the Endogenous Thrombin Potential obtained when spiking patient's plasma with Factor IX concentrates to that obtained when spiking patient's plasma with recombinant porcine FVIII on emicizumab prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Maissa Janbain, MD, MS, Principal Investigator — Tulane University
Locations (2):
- United States (2):
  - Tulane University Lakeside Hospital and Clinics, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: Undecided